CLINICAL TRIAL: NCT04908839
Title: Validation of the French Version of the Stapesplasty Outcome Test 25 (SPOT-25)
Acronym: QOLOTOSC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MDL _2021_12
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Otosclerosis
Keywords: SPOT-25
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- case: patient with otosclerosis: Diagnosis of otosclerosis with indication for primary stapedial surgery by the combination of arguments
  Interventions: Other: spot-25 questionnaire
- case: otosclerosis patient with surgery: otosclerosis patient with surgery
  Interventions: Other: spot-25 questionnaire
- controle: Absence of known otological pathology: Absence of known otological pathology
  Interventions: Other: spot-25 questionnaire

INTERVENTIONS:
Other: spot-25 questionnaire — spot-25 questionnaire

SUMMARY:
Inclusion (J0):

* Audiometry (as part of the treatment, only for cases)
* Clinical evaluation (within the framework of care, only for cases)
* Passage of the French version of the SPOT-25 questionnaire

Visit 1 (D0 + 3 ± 1 week): only for cases Second examination of the French version of the SPOT-25 questionnaire (re-test) either by telephone and e-mail, or during a consultation or hospitalization, if this occurs within a compatible time frame.

Visit 2 (3-6 months postoperatively): only for operated patients Third examination of the French version of the SPOT-25 questionnaire either by telephone and e-mail, or during a consultation or hospitalization, if this occurs within a compatible time frame.

DETAILED DESCRIPTION:
Inclusion (J0):

* Audiometry (as part of the treatment, only for cases)
* Clinical evaluation (within the framework of care, only for cases)
* Passage of the French version of the SPOT-25 questionnaire

Visit 1 (D0 + 3 ± 1 week): only for cases Second examination of the French version of the SPOT-25 questionnaire (re-test) either by telephone and e-mail, or during a consultation or hospitalization, if this occurs within a compatible time frame.

Visit 2 (3-6 months postoperatively): only for operated patients Third examination of the French version of the SPOT-25 questionnaire either by telephone and e-mail, or during a consultation or hospitalization, if this occurs within a compatible time frame.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged> 18 years
* Diagnosis of otosclerosis with indication for primary stapes surgery by the combination of the arguments:

  * Clinical: normal eardrum and audiometry revealing conductive or mixed hearing loss with audiometric Rinne of> 15 dB and absence of stapedial reflex.
  * Radiological: otosclerotic foci on preoperative CT scan
* Non-opposition to participating in the study
* Good understanding of French
* Affiliate or beneficiary of a health insurance plan

Inclusion criteria for witnesses:

* Person aged> 18 years
* Absence of known otological pathology
* Without otological surgical history
* Non-opposition to participating in the study
* Good understanding of French

Exclusion Criteria:

* Comorbidity that may interfere with the interpretation of results
* History of stapes surgery
* Person benefiting from a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with otosclerosis and person with a known Absence of otological pathology
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the total score of cases and controls for the French version of the SPOT-25 questionnaire | 1 DAY
  The SPOT-25 questionnaire includes 25 items and can be divided into 4 subscores: hearing function (items 1-10), tinnitus (items 11-13), mental condition (items 14-19), and social restrictions (items 20-24). In addition, 1 item focuses on the general evaluation of the impact of otosclerosis on HRQOL (item 25). Each question needs to be rated on a six-point ordinal scale from 0 (i.e., no impact) to 5 (i.e., most severe impact), depending on the level of inconvenience or frequency of symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Fondation Adolphe de Rothschild, Paris
  - Amélie YAvchitz, Paris, Île-de-France Region